CLINICAL TRIAL: NCT06511466
Title: Evaluation of a Training Model for the Proficient Use of the Belmont Rapid Infuser
Brief Title: Belmont Rapid Infuser Education
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: BRI
Record Dates: First submitted 2013-08-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia
Keywords: Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Belmont Rapid Infuser (BRI) represents medical equipment with potential to elicit serious injury. The device is used infrequently and at irregular time of day which makes training and competency of operation difficult to ensure. In the investigators institution BRI is used infrequently, usually for pediatric trauma cases and liver transplant cases.

The current teaching module for BRI includes oral slide presentation and live demonstration of BRI assembly and a written test. The effectiveness of this module has never been tested. The investigators central hypothesis is that modified training will significantly increase proficiency rate. The current traditional teaching module is insufficient to retain knowledge and be proficient. The investigators plan to study the current teaching module (traditional test method) to evaluate its effectiveness in acquisition of proficiency and retention of knowledge and skills.

The aims of this study are:

Aim 1. To evaluate the current method of teaching on proficient use of the BRI, Hypothesis: The use of traditional test method is not effective as less than 50% will pass in the first attempt.

Aim 2. Re-design the teaching module if necessary to optimize the method if the current method is found to be inadequate Hypothesis: Restructured test that provides a hand-on training as opposed to only an oral presentation with the traditional test will be associated with a higher pass rate (>80%).

Aim 3. To perform the success with BRI assembly in clinician pairs versus a single clinician.

Hypothesis: Working in pairs is better than working as a single person in setting up the BRI within the recommended time limit.

Aim 4: To better define proficiency with the use of the BRI with respect to retention of knowledge and skills after initial teaching and successful tests.

Hypothesis: Retention at 3 months is required irrespective of the initial training method in order to retain competency. Retention at 3 months will be higher with the restructured training than with the traditional training method.

The investigators will employ a quality improvement methodology invoking a PDSA (Plan-Do-Study Act) ramp to evaluate and improve the training model as necessary.

JHACO requires that all equipment users be trained annually in proper operating procedures for the equipment they use and that the training is documented. The investigators propose that retraining may have to be done more frequently in order to retain knowledge especially when this knowledge is to be used during emergency care of children.

Medical equipment in the OR may be divided into 4 categories based on the frequency of use and risk of injury. BRI belongs to the category of low frequency of use, but high risk of injury. These categories of medical equipment will require different strategies for teaching and training that need to be explored.

If the investigators current teaching module is found to be an effective one, it could be replicated for other types of medical equipment as well as spread to other institutions that use similar equipment.

DETAILED DESCRIPTION:
This study is a randomized non-blinded study. Since the investigators are following a quality improvement methodology, there is only an intervention group and not a control group. All participants will receive the training intervention.

Study participants for phase 1 will include subjects in each of following categories: faculty, certified registered nurse anesthetists (CRNA), Registered Nurses and pediatric anesthesia fellows. Participants will be recruited from the Department of Anesthesia with no attention to gender, race, age, or socioeconomic status.

Participants will be tested with the traditional test method as a first step. Based on the outcomes of this test method, a decision would be made to conduct the restructured training. Traditional method is the current method used which involves oral slide presentation followed by demonstration and written test. There will be a video presentation followed by a demonstration by and experienced Anesthesia Tech Restructured training that the investigators are proposing will consist of an oral slide presentation and will follow hands-on assembly and written test. The 'hands-on assembly' will be the new training technique that will be different from the original technique.

ELIGIBILITY:
Study participants for phase 1 will include subjects in each of following categories: faculty, certified registered nurse anesthetists (CRNA), Registered Nurses and pediatric anesthesia fellows. Participants will be recruited from the Department of Anesthesia with no attention to gender, race, age, or socioeconomic status. -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesia Faculty, Fellows and CRNA's
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Proficiency | July 2013
  Primary outcome: proficiency: composite score of pass - pass on BRI assembly and pass on knowledge test.

SECONDARY OUTCOMES:
Retention | June 2014
  Retention of proficiency at 3 months after delivery of the effective teaching module.